CLINICAL TRIAL: NCT03517826
Title: Validity and Reliability of The Turkish Version of Breathlessness Beliefs
Brief Title: Validity and Reliability of The Turkish Version of Breathlessness Beliefs Questionnaire
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Seda Saka, MSc, PT, Bezmialem Vakif University
Other Study IDs: bvussaka02
Record Dates: First submitted 2018-04-25; First posted 2018-05-07 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Dyspnea; COPD
Keywords: COPD; Dyspnea; Kinesiophobia
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, we aimed to evaluate the validity and reliability of the Turkish version of the Breathlessness Beliefs Questionnaire-BBQ in our study.

DETAILED DESCRIPTION:
Pulmonary diseases are a common cause of mortality and morbidity throughout the world. In pulmonary diseases such as asthma and COPD, the main symptom is dyspnea and it causes activity limitation. Dyspnea is defined as the difficulty that a person experiences during breathing. As a result of painful situations or injuries, avoidance of physical activity or movement due to the fear of repetition of the problem are defined as kinesophobia. Pulmonary patients are compensated by reducing the rate of activity, while avoiding dyspnea.This reduces the severity of the symptom that precedes the symptom that may occur. As a result, dyspnea causes kinesyphobia. Decrease in the level of activity; social isolation, fear of dyspnea, depression and anxiety result in a stubborn cycle, quality of life is reduced. The Breathlessness Beliefs Questionnaire (BBQ) was developed based on the Tampa Kinesiophobia Scale to assess dyspnea and dyspnoea-related kinesophobia and anxiety in respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC<%70
* To be able to read and understand Turkish

Exclusion Criteria:

* Having undergone a COPD exacerbation in the last 6 weeks
* Having comorbidities affecting ambulance
* Having cognitive disorders

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Breathlessness Beliefs Questionnaire-BBQ | 3 Minutes
  Breathlessness Beliefs Questionnaire-BBQ Breathlessness Perception Questionnaire; is a measure evaluating kinesophobia and anxiety due to the breathlessness of 17 questions answered by one's own practice. Patients score from 1 to 5 (I strongly agree). High scores indicate high levels of kinesiophobia and anxiety due to breathlessness.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, MSc, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] De Peuter S, Janssens T, Van Diest I, Stans L, Troosters T, Decramer M, Van den Bergh O, Vlaeyen JW. Dyspnea-related anxiety: The Dutch version of the Breathlessness Beliefs Questionnaire. Chron Respir Dis. 2011;8(1):11-9. doi: 10.1177/1479972310383592. Epub 2010 Dec 20. PMID 21172990
- [Result] Wu Q, Guo A, Zhao Y, Li S, Huang H. Reliability and validity of the Chinese version of the Breathlessness Beliefs Questionnaire. Chron Respir Dis. 2018 May;15(2):114-122. doi: 10.1177/1479972317715551. Epub 2017 Jun 21. PMID 28635313